CLINICAL TRIAL: NCT01055769
Title: An Open Label, Single Dose, 2-Way, Randomized Cross-Over Bioequivalence Study Comparing Linezolid 600 Mg Oral Suspension With 600 Mg Tablet In Chinese Healthy Male Subjects
Brief Title: Bioequivalence Study Comparing Linezolid 600 Mg Oral Suspension With 600 Mg Tablet In Chinese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A5951152
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Volunteers
Keywords: Bio-equivalence; Linezolid OS; Linezolid tablet
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Subjects will accept Linezolid OS 600 MG first, after 4 days wash-out, then will accept Linezolid tablet 600 MG.
  Interventions: Drug: Linezolid
- Group 2 (Other): Subjects will accept Linezolid tablet 600 MG first, after 4 days wash-out, then will accept Linezolid OS 600 MG.
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — 1. Linezolid OS 600 MG
  2. Linezolid Tablet 600 MG
  Other Names: Zyvox
  Arms: Group 1
Drug: Linezolid — 1. Linezolid Tablet 600 MG
  2. Linezolid OS 600 MG
  Other Names: Zyvox
  Arms: Group 2

SUMMARY:
The purpose of this study is to estimate the bioequivalence comparing Linezolid 600 MG Oral Suspension with 600 MG tablet in Chinese healthy male subjects. This study data will be used to support Linezolid OS NDA in China.

DETAILED DESCRIPTION:
To support Linezolid NDA in China.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* 18-40 years old, male.
* BMI 19-24kg/m2.

Exclusion Criteria:

* Alcohol, drug, smoke user.
* Sensitive to oxazolidinones antibiotics class drug or heparin.
* Severe medical or psychiatric condition or laboratory abnormality.
* Blood donation.
* 12-ECG abnormal.
* Treatment with study drug; clinically significant.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Shanghai, China

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951152&StudyName=Bioequivalence%20Study%20Comparing%20Linezolid%20600%20Mg%20Oral%20Suspension%20With%20600%20Mg%20Tablet%20In%20Chinese%20Healthy%20Male%20Subjects

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a single site in China.
Groups:
- Linezolid 600 mg Oral Suspension, Then Linezolid 600 mg Tablet: Linezolid oral suspension 600 mg once in morning (at approximately 8:00 AM, after fasting overnight) on Day 1 in first intervention period and Linezolid tablet 600 mg once in morning (at approximately 8:00 AM, after fasting overnight) on Day 1 in second intervention period (after washout period).
- Linezolid 600 mg Tablet, Then Linezolid 600 mg Oral Suspension: Linezolid tablet 600 mg once in morning (at approximately 8:00 AM, after fasting overnight) on Day 1 in first intervention period and Linezolid oral suspension 600 mg once in morning (at approximately 8:00 AM, after fasting overnight) on Day 1 in second intervention period (after washout period).
Period: First Intervention
Arm/Group | Linezolid 600 mg Oral Suspension, Then Linezolid 600 mg Tablet | Linezolid 600 mg Tablet, Then Linezolid 600 mg Oral Suspension
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period of Atleast 4 Days
Arm/Group | Linezolid 600 mg Oral Suspension, Then Linezolid 600 mg Tablet | Linezolid 600 mg Tablet, Then Linezolid 600 mg Oral Suspension
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Linezolid 600 mg Oral Suspension, Then Linezolid 600 mg Tablet | Linezolid 600 mg Tablet, Then Linezolid 600 mg Oral Suspension
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Linezolid: Linezolid 600 mg once (oral suspension or tablet) in morning (at approximately 8:00 AM) on Day 1 after fasting overnight.
Arm/Group | Linezolid
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: Years] | 25.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time curve from time zero (pre-dose) to the time of the last measurable concentration (AUClast).
Time Frame: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: Pharmacokinetic concentration population: all randomized and treated participants who had at least 1 concentration in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: microgram*hour/milliliter (mcg*h/mL)
Groups:
- Linezolid 600 mg Oral Suspension: Linezolid oral suspension 600 mg once in morning (at approximately 8:00 AM) on Day 1 after fasting overnight.
- Linezolid 600 mg Tablet: Linezolid tablet 600 mg once in morning (at approximately 8:00 AM) on Day 1 after fasting overnight.
Arm/Group | Linezolid 600 mg Oral Suspension | Linezolid 600 mg Tablet
Number analyzed (Participants) | 20 | 20
microgram*hour/milliliter (mcg*h/mL) | 108.90 (21.66) | 112.00 (24.74)
Statistical Analysis 1: Comparison: Linezolid 600 mg Oral Suspension vs Linezolid 600 mg Tablet; Natural log transformed AUClast of linezolid was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Linezolid 600 mg oral suspension was the Test treatment, while linezolid 600 mg tablet was the Reference treatment; Adjusted Geometric Means Ratio = 97.81, 90% CI 2-sided [93.11 to 102.75]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration within the dosing interval was directly obtained from the concentration-time data.
Time Frame: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Linezolid 600 mg Oral Suspension | Linezolid 600 mg Tablet
Number analyzed (Participants) | 20 | 20
microgram/milliliter (mcg/mL) | 15.51 (3.53) | 13.68 (3.53)
Statistical Analysis 1: Comparison: Linezolid 600 mg Oral Suspension vs Linezolid 600 mg Tablet; Natural log transformed Cmax of linezolid was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Means Ratio = 113.67, 90% CI 2-sided [105.26 to 122.75]

3. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)]
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Linezolid 600 mg Oral Suspension | Linezolid 600 mg Tablet
Number analyzed (Participants) | 20 | 20
mcg*h/mL | 109.20 (21.72) | 112.60 (24.94)
Statistical Analysis 1: Comparison: Linezolid 600 mg Oral Suspension vs Linezolid 600 mg Tablet; Natural log transformed AUCinf of linezolid was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric means ratio = 97.65, 90% CI 2-sided [92.92 to 102.63]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: The time of the first occurrence of peak concentration observed directly from data.
Time Frame: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Linezolid 600mg Tablet: Linezolid tablet 600 mg once in morning (at approximately 8:00 AM) on Day 1 after fasting overnight.
Arm/Group | Linezolid 600 mg Oral Suspension | Linezolid 600mg Tablet
Number analyzed (Participants) | 20 | 20
hours | 0.63 [0.50 to 2.00] | 1.50 [0.50 to 4.00]

5. Secondary Outcome: Terminal Half-Life (t1/2)
Description: Plasma terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Linezolid 600 mg Oral Suspension | Linezolid 600 mg Tablet
Number analyzed (Participants) | 20 | 20
hours | 5.08 (0.70) | 5.13 (0.92)

ADVERSE EVENTS:
Time Frame: Baseline to Day 3
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid 600 mg Oral Suspension | Linezolid 600 mg Tablet
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid 600 mg Oral Suspension (N=20) | Linezolid 600 mg Tablet (N=20)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.